CLINICAL TRIAL: NCT06038357
Title: Evaluation of "Cognitive Behavioral Intervention for Trauma in Schools" (CBITS) in Child Welfare Programs in Germany: A Randomized Controlled Trial
Brief Title: CBITS - Treat Trauma in Child Welfare
Acronym: CBITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Ulm (Other)
Collaborators: Ruhr University of Bochum (Other); Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dr. Elisa Pfeiffer, Principal Investigator (Chief Psychologist), University Hospital Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFG PF 990/4-1 - AO 692822
Record Dates: First submitted 2023-07-24; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: children; adolescents; PTSD; trauma-focused group intervention; randomized controlled trial; child welfare programs; CBITS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Schools

STUDY DESIGN:
Intervention Model Description: CBITS intervention vs. Treatment as Usual (TAU+)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBITS (Experimental): Cognitive Behavioral Intervention for Trauma in Schools (CBITS)
  Interventions: Behavioral: CBITS
- Treatment as usual (TAU+) (Active Comparator): Enhanced Treatment as Usual means regular care in child welfare program and mental health care. They also receive feedback on their assessments and a treatment recommendation.
  Interventions: Other: TAU+

INTERVENTIONS:
Behavioral: CBITS — The CBITS program is a skills-based group and individual intervention, which uses evidence-based cognitive-behavioral techniques (e.g. psychoeducation, relaxation, social problem solving, cognitive restructuring, and exposure) and is designed for delivery by mental health professionals. The program consists of 10 45-minute group sessions (about 6-8 students/participants per group), 1-3 individual sessions, 2 parent/caregiver psychoeducational sessions, and 1 teacher/ child welfare staff educational session. For this study, we will specifically train and supervise study therapists to deliver the intervention within child welfare programs.
  Other Names: Cognitive Behavioral Intervention for Trauma in Schools
  Arms: CBITS
Other: TAU+ — In the control condition (TAU+), child welfare programs will follow their usual procedures (i.e. routine care of child welfare, referral to medical practitioners and psychotherapists, handling of prescribed medication, referral to inpatient treatments in case of risk to self and others) which reflects treatment as usual in child welfare programs and the mental health care system in Germany. Additionally, participants in the control condition will receive the same baseline assessment and reporting of screening results as participants in the treatment condition after each assessment.
  Arms: Treatment as usual (TAU+)

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of the trauma-focused group intervention CBITS compared with enhanced treatment as usual (TAU+) in child welfare programs in Germany. The target group are traumatized children and adolescents in out-of-home care who report posttraumatic stress symptoms (PTSS).

DETAILED DESCRIPTION:
The study objectives are

1. Evaluate the effectiveness of CBITS compared to TAU+ regarding PTSS symptom reduction (primary outcome), anxiety, depression, quality of life and functional level, and continuance of the child welfare program (secondary outcomes) at 4-month follow-up
2. Investigate potential long-term effects of the treatment in the CBITS condition regarding the primary and secondary outcomes at 10-month follow-up.
3. Implement CBITS as an outreach intervention into routine mental health care for traumatized children, to evaluate treatment fidelity, treatment completion and investigate different potential individual or structural factors that might have an impact on the implementation.
4. To assess the readiness in child welfare programs to collaborate with mental health services and the role of institutional environments for developmental trajectories.

Participants and their caregivers will complete questionnaires at three measurement time points. Weekly PTSS symptom monitoring during treatment and alliance ratings (participants and therapists) at the beginning and the end of the intervention will be implemented. Trained therapists at three study centers (Marburg, Ulm, Bochum) will complete questionnaires before their training and after CBITS implementation. Site monitoring and auditing, as well as reliability checks of the data will be conducted by an independent data manager. Randomization will be implemented by an independent Institute at Ulm University. Standard Operating Procedures (SOPs) to address patient recruitment, data collection, data management, reporting for adverse events, and change management will be provided. Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect were performed via the program G-Power, in collaboration with an independent statistical advisor, before proposal submission. A plan for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results are prepared in collaboration with the independent statistical advisor. We will following Intention-to-treat (ITT) principles in our analyses. The statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, are specified in the study protocol which will be published before data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-16 years, because this age range reflects the age range in the CBITS evaluation studies, and this age range is specified in the CBITS manual and toolkit).
2. Having experienced at least one traumatic event (based on DSM-5 or ICD-10/ICD-11 criteria) as CBITS is designed for children and adolescents with a trauma history.
3. At least moderate PTSS (at least 21 points on the CATS-2) as this is recommended in the intervention manual. Participants don't have to fulfill PTSD criteria as the manual does not name this a pre-condition for participation. Additionally, there is large evidence that also youth with subthreshold PTSS show high functional impairment, but respond very well to trauma-focused interventions.
4. Being currently cared for by a child welfare program (safe and stable living conditions), planned further stay in the program for at least 12 months in order to complete the CBITS intervention and 10-month follow-up.
5. Willingness and informed assent/consent of the participant as well as informed consent of the caregiver/legal guardian to participate in the study (sufficient motivation for group intervention and compliance with the study design).

Exclusion Criteria:

1. Current psychosis for safety reasons and in because in this case another intervention another intervention has priority (same explanation for 2-4).
2. severe harm to self or others
3. severe substance disorder
4. acute suicidality
5. Severe mental retardation as there is a certain necessity of sufficient cognitive abilities to benefit from CBITS, to recall trauma memories and to create a trauma narrative.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen - Second Version (CATS-2 self-report) | baseline, 4-month follow-up, 10-month follow-up (primary endpoint 4-months follow up)
  The CATS-2 is a questionnaire to screen for potentially traumatic events and assesses symptoms of PTSD/Complex-PTSD (CPTSD) (according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and International Classification of Diseases Version 11 (ICD-11)) in children and adolescents. The minimal score value is "0", the maximum score value is "60", while higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS) (self-and caregiver report) | baseline, 4-month follow-up, 10-month follow-up
  The RCADS is a 47-item, self- and caregiver-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). For the anxiety subscale the minimum score value is "0", the maximum score value is "111", while higher scores mean more anxiety. For the depression subscale the minimum score value is "0", the maximum score value is "30", while higher scores mean worse depressive symptoms. Therefore, the minimum score value is "0", the maximum score value is "141", while higher scores mean a worse outcome.
Screening and Promotion of Children and Adolescents Health: A European Public Health Perspective (KIDSCREEN questionnaire) (self-and caregiver report) | baseline, 4-month follow-up, 10-month follow-up
  Quality of life will be assessed via the KIDSCREEN-10 which is a generic health related quality of life measure. The minimum score value is "10", the maximum score value is "50", while higher scores mean a better quality of life.
Child and Adolescent Trauma Screen - Second Version (CATS-2 caregiver-report) | baseline, 4-month follow-up, 10-month follow-up
  corresponding measure to CATS-2 self-report, completed by the participants' caregivers. The minimum score value is "0", the maximum score value is "60", while higher scores mean a worse outcome.
Children's Global Assessment Scale (CGAS Caregiver-report) | baseline, 4-month follow-up, 10-month follow-up
  The level of functioning will be assessed via the CGAS. The minimum score value is "1", the maximum score value is "100", while higher scores mean a higher functioning level.

OTHER OUTCOMES:
Non-standardized quantitative questionnaire to collect study feedback | 4-month follow-up, 10-month follow-up
  Via a non-standardized quantitative questionnaire, participants, caregivers, and therapists will be asked about their experiences with the overall study and the CBITS intervention. The questionnaire for participants consists of 13 Items. The minimum score value is "0", the maximum score value is "65". A higher score means a better Feedback. The questionnaire for the caregivers consists of 9 Items. 7 of them can be rated on a Likert-Scale. The minimum score value is "7", the maximum score value is "42". Higher scores mean a worse feedback. The questionnaire for the therapists consists of 19 Items. 6 can be rated on a Likert-Scale. The minimum score value is "6", the maximum score value is "36", while higher scores mean a worse feedback.
Non-standardized qualitative interview to collect study feedback | 4-month follow-up, 10-month follow-up
  Via non-standardized qualitative interview using 13 items the participants, caregivers and therapists will be asked about their overall experiences during the study and the CBITS intervention.
Child and Adolescent Mental Health Service Receipt Inventory - German (CAMHSRI-German caregiver-report) | baseline, 4-month follow-up, 10-month follow-up
  Use of medical, psychosocial and child welfare services in both conditions will be assessed in a standardized manner by the CAMHSRI-DE. Completed by the caregivers.
Implementation Climate Scale (ICS Caregiver-report) | baseline
  The ICS is an 18-item questionnaire measuring the degree to which the organizational climate is supportive of evidence-based practice (EBP) implementation. The items form six subscales including focus on EBP, educational support for EBP, recognition for EBP, rewards for EBP, selection for EBP and selection for openness. The minimum score value for every subscale and in total is "0", the maximum score value is "4", while higher scores indicate a better fit of the intervention in the environment.
Evidence-Based Practice Attitude Scale (EBPAS-36 Caregiver-report) | baseline
  The EBPAS-36 is a 36-item questionnaire assessing attitudes of mental health providers towards the adoption of EBP. The items form 12 subscales (requirements, appeal, openness, divergence, limitations, fit, monitoring, balance, burden, job security, organizational support, feedback). The minimum score value for every subscale and in total is "0", the maximum score value is "4", while higher scores indicate a better attitude towards evidence-based practice.
CBITS original adherence and fidelity measure | through study completion, an average of 10 weeks
  The therapist adherence and fidelity will be assessed by the CBITS Adherence/Fidelity measure which is a 4 Item scale. The minimum score value is "0", the maximum is "3", while higher scores mean that the topic has been thoroughly covered.
Child and Adolescent Trauma Screen - Second and Short Version (CATS-2 self-report) | through study completion, an average of 10 weeks
  At the beginning of every CBITS session, the participants complete a short version of the CATS-2 symptom screener. The minimum score value is "0", the maximum score value is "21", while higher scores mean a worse outcome.
Therapeutic Alliance Scales for Children - Revised (TASC-r) | through study completion, an average of 10 weeks
  The working alliance between therapists and participants will be assessed via TASC-r (questions on therapist and group alliance). The measure will be completed by the participants and therapists. The minimum score value is "0", the maximum score value is "4", while higher scores mean a better outcome.
Inventory for the Assessment of Negative Effects of Psychotherapy for children and adolescents (Children-INEP) (self-and caregiver report) | 4-month follow-up, 10-month follow-up
  The Children-INEP is an 18-item questionnaire (12 items on subscale "negative effects" and 6 items on subscale "unethical behavior and malpractice") which assesses unwanted side effects in psychotherapy after several months post-treatment via self-and care-giver report. The minimum score value for the subscale negative effects is "0", the maximum score values is "12", while higher rates mean more negative side effects. The items for the subscale unethical behavior and malpractice will be rated on individual item level with a minimum score value of "1" and maximum score value of "4" for each item. Higher scores are worse therapeutic behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Pfeiffer, PhD, Principal Investigator — Ulm University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Yes - Individual participant data (IPD) will be made available to other researchers on request, after publication of the main results and after data sharing agreements are concluded. All IPD that underlie results in a publication will be shared. The study protocol and statistical analysis plan will be shared. IPD and additional supporting information will become available for 2 years once summary data is published. Requests for IPD data and additional supporting information will be reviewed by the leaders of the project (E. Pfeiffer and C. Sachses). There is no web address about the plan to share IPD available.

REFERENCES:
- [Background] Sachser C, Berliner L, Risch E, Rosner R, Birkeland MS, Eilers R, Hafstad GS, Pfeiffer E, Plener PL, Jensen TK. The child and Adolescent Trauma Screen 2 (CATS-2) - validation of an instrument to measure DSM-5 and ICD-11 PTSD and complex PTSD in children and adolescents. Eur J Psychotraumatol. 2022 Aug 1;13(2):2105580. doi: 10.1080/20008066.2022.2105580. eCollection 2022. PMID 35928521
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Waldmann T, Stiawa M, Dinc U, Saglam G, Busmann M, Daubmann A, Adema B, Wegscheider K, Wiegand-Grefe S, Kilian R. Costs of health and social services use in children of parents with mental illness. Child Adolesc Psychiatry Ment Health. 2021 Feb 20;15(1):10. doi: 10.1186/s13034-021-00360-y. PMID 33610177
- [Background] Ehrhart MG, Aarons GA, Farahnak LR. Going above and beyond for implementation: the development and validity testing of the Implementation Citizenship Behavior Scale (ICBS). Implement Sci. 2015 May 7;10:65. doi: 10.1186/s13012-015-0255-8. PMID 25948489
- [Background] Rye M, Torres EM, Friborg O, Skre I, Aarons GA. The Evidence-based Practice Attitude Scale-36 (EBPAS-36): a brief and pragmatic measure of attitudes to evidence-based practice validated in US and Norwegian samples. Implement Sci. 2017 Apr 4;12(1):44. doi: 10.1186/s13012-017-0573-0. PMID 28372587
- [Background] Bieda A, Pflug V, Scholten S, Lippert MW, Ladwig I, Nestoriuc Y, Schneider S. [Unwanted Side Effects in Children and Youth Psychotherapy - Introduction and Recommendations]. Psychother Psychosom Med Psychol. 2018 Sep;68(9-10):383-390. doi: 10.1055/s-0044-102291. Epub 2018 May 30. German. PMID 29847849
- [Derived] Pfeiffer E, Dorrie L, Koksal J, Krech F, Muche R, Segler J, Sachser C. Evaluation of "Cognitive Behavioral Intervention for Trauma in Schools" (CBITS) in child welfare programs in Germany: study protocol of a randomized controlled trial. Trials. 2024 Jun 19;25(1):399. doi: 10.1186/s13063-024-08190-x. PMID 38898537